CLINICAL TRIAL: NCT01678976
Title: Tolerability and Pharmacokinetics of a Single 900 mg Oral Dose of BIA 2-093 and Oxcarbazepine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-104
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; Epilepsy; Oxcarbazepine
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 BIA 2-093 + Oxcarbazepine (Experimental): Period 1 - Subjects recieved 900 mg of BIA 2-093 Period 2 - Subjects recieved 900 mg of oxcarbazepine
  Interventions: Drug: BIA 2-093; Drug: Oxcarbazepine
- Group 2 Oxcarbazepine + BIA 2-093 (Active Comparator): Period 1 - Subjects recieved 900 mg of oxcarbazepine Period 2 - Subjects recieved 900 mg of BIA 2-093
  Interventions: Drug: BIA 2-093; Drug: Oxcarbazepine

INTERVENTIONS:
Drug: BIA 2-093 — Tablets containing BIA 2-093 in doses of 300 and 600 mg
  Other Names: Eslicarbazepine acetate
Drug: Oxcarbazepine — Tablets containing 300 mg and 600 mg of Trileptal®
  Other Names: Trileptal®

SUMMARY:
To investigate the pharmacokinetics of a single 900 mg oral dose of BIA 2-093 and a single 900 mg oral dose of Oxcarbazepine in healthy volunteers and to assess the tolerability of a single 900 mg dose of BIA 2-093 and Oxcarbazepine.

DETAILED DESCRIPTION:
Single centre, open label, balanced randomised, two-way crossover study in 12 healthy volunteers. The study consisted of 2 periods separated by a washout period of 7 days or more. On each of the study periods the volunteers received either a single 900 mg oral dose of BIA 2-093 or a single 900 mg oral dose of Oxcarbazepine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests acceptable.
* Subjects who were negative for HBs Ag, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* In case of female volunteers, subjects who were not of childbearing potential by reason of surgery or, if of childbearing potential, used one of the following methods of contraception: double-barrier, intrauterine device or abstinence.
* In case of female volunteers, subjects who had a negative pregnancy test at screening and admission

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used over-the-counter medication excluding oral routine vitamins but including mega dose vitamin therapy within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 2 months of their first admission.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated and/or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* In case of female volunteers, subjects who were pregnant or breast-feeding.
* In case of female volunteers, subjects who were of childbearing potential and did not use an approved effective contraceptive method or used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2002-03; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, MD, PhD, Principal Investigator — BIAL - Portela & Cª S.A
Locations (1):
- BIAL - Portela & Cª - Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Trofa, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1 - BIA 2-093; Period 2 - Oxcarbazepine: Period 1 - Subjects recieved 900 mg of BIA 2-093 Period 2 - Subjects recieved 900 mg of oxcarbazepine
- Period 1 - Oxcarbazepine; Period 2 - BIA 2-093: Period 1 - Subjects recieved 900 mg of oxcarbazepine Period 2 - Subjects recieved 900 mg of BIA 2-093
Period: First Period
Arm/Group | Period 1 - BIA 2-093; Period 2 - Oxcarbazepine | Period 1 - Oxcarbazepine; Period 2 - BIA 2-093
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Period: Second Period
Arm/Group | Period 1 - BIA 2-093; Period 2 - Oxcarbazepine | Period 1 - Oxcarbazepine; Period 2 - BIA 2-093
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1 - BIA 2-093; Period 2 - Oxcarbazepine | Period 1 - Oxcarbazepine; Period 2 - BIA 2-093 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) was acessed for BIA 2-093 metabolites (BIA 2-194; BIA 2-195) and Oxcarbazepine.
Time Frame: at pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Population: Values are described for single dose of BIA 2-093 or oxcarbazepine respectively for Group 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 900 mg od: BIA 2-093, ESL Eslicarbazepine acetate
- Oxcarbazepine 900 mg od: Oxcarbazepine, Trileptal®
Arm/Group | BIA 2-093 900 mg od | Oxcarbazepine 900 mg od
Number analyzed (Participants) | 6 | 6
ng/mL
  Cmax (BIA 2-194) | 15753 (3781) | 5978 (1136)
  Cmax (BIA 2-195) | 428 (88.6) | 1708 (751)
  Cmax (Oxcarbazepine) | 140 (37.7) | 1268 (656)

2. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Area under the plasma concentration versus time curve (AUC) to last measurable time point (AUC0-t) was acessed for BIA 2-093 metabolites (BIA 2-194; BIA 2-195) and Oxcarbazepine.
Time Frame: at pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Population: Values are described for single dose of BIA 2-093 or oxcarbazepine respectively for Group 1 and 2.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- BIA 2-093 900 mg od: BIA 2-093, ESL, Eslicarbazepine acetate
Arm/Group | BIA 2-093 900 mg od | Oxcarbazepine 900 mg od
Number analyzed (Participants) | 6 | 6
ng*h/mL
  AUC0-t (BIA 2-194) | 299065 (65077) | 214433 (45162)
  AUC0-t (BIA 2-195) | 13877 (2867) | 49124 (18926)
  AUC0-t (Oxcarbazepine) | 1821 (693) | 6549 (3927)

3. Other Pre Specified Outcome: Total of Subjects Reporting at Least One Adverse Event
Description: Monitoring of Adverse Events throughout the study: Safety was evaluated from the number of reported adverse events (AEs) by patient
Time Frame: 4 weeks
Measure: Number; unit: subjects reporting at least 1 AE
Groups:
- BIA 2-093: BIA 2-093, ESL, Eslicarbazepine
- Oxcarbazepine: Oxcarbazepine, Trileptal
Arm/Group | BIA 2-093 | Oxcarbazepine
Number analyzed (Participants) | 12 | 13
subjects reporting at least 1 AE
  All treatment-emergent AEs | 6 | 6
  Possibly related to treatment AEs | 5 | 4

ADVERSE EVENTS:
Arm/Group | BIA 2-093 | Oxcarbazepine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 10/12 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 (N=12) | Oxcarbazepine (N=13)
Dizziness (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 1 | 2
Concentration impairment (Nervous system disorders) | 2 | 0
Lipothymia (Nervous system disorders) | 1 | 0
Nystagmus NOS (Nervous system disorders) | 2 | 0
Parasthesiae circumoral (Nervous system disorders) | 2 | 0
Taste bitter (Nervous system disorders) | 2 | 0
Thinking reduced (Nervous system disorders) | 0 | 2
Syncope vasovagal (Nervous system disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Application site bruise (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Venipuncture site bruise (General disorders) | 1 | 0
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sensation of pressure in ear (Ear and labyrinth disorders) | 0 | 2
CPK increased (Investigations) | 0 | 1
Nodule subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes